CLINICAL TRIAL: NCT02292719
Title: A Randomized, Open-Label Study to Evaluate the Safety and Efficacy of the Co-Administration of Ombitasvir/ABT-450/Ritonavir (Ombitasvir/ABT-450/r) With Sofosbuvir (SOF) With or Without Ribavirin (RBV) in Subjects With Genotype 2 Chronic Hepatitis C Virus (HCV) Infection or Genotype 3 HCV Infection With or Without Cirrhosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Ombitasvir/ABT-450/Ritonavir With Sofosbuvir With or Without Ribavirin in Adults With Chronic Hepatitis C Virus Infection
Acronym: Quartz II/III
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-567; 2014-003147-35 (EudraCT Number)
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Hepatitis C Virus; Genotype 2; Chronic Hepatitis C; Genotype 3; Non-cirrhotic; Cirrhotic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ombitasvir; paritaprevir; Ritonavir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm A (genotype [GT]3, noncirrhotic) (Experimental): Ombitasvir (OBV)/paritaprevir (PTV)/ritonavir (r) 25/150/100 mg once daily (QD) and sofosbuvir (SOF) 400 mg QD for 12 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir
- Arm B (GT3, noncirrhotic) (Experimental): OBV/PTV/r (25/150/100) mg QD with SOF (400 mg QD) and ribavirin (RBV; weight-based 1,000 mg or 1,200 mg daily divided twice daily [BID]) for 12 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir; Drug: Ribavirin (RBV)
- Arm C (GT2, noncirrhotic) (Experimental): OBV/PTV/r (25/150/100) mg QD with SOF (400 mg QD) and RBV (weight- based 1,000 mg or 1,200 mg daily divided BID) for 8 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir; Drug: Ribavirin (RBV)
- Arm D (GT2, noncirrhotic) (Experimental): OBV/PTV/r (25/150/100) mg QD with SOF (400 mg QD) and RBV (weight-based 1,000 mg or 1,200 mg daily divided BID) for 6 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir; Drug: Ribavirin (RBV)
- Arm E (GT3, cirrhotic) (Experimental): OBV/PTV/r (25/150/100) mg QD with SOF (400 mg QD) and RBV (weight-based 1,000 mg or 1,200 mg daily divided BID) for 12 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir; Drug: Ribavirin (RBV)
- Arm F (GT3, noncirrhotic) (Experimental): OBV/PTV/r (25/150/100) mg QD and SOF (400 mg QD) for 12 weeks.
  Interventions: Drug: OBV/PTV/r; Drug: Sofosbuvir

INTERVENTIONS:
Drug: OBV/PTV/r — Tablet
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ritonavir (r) also known as Norvir; VIEKIRAX combination tablets; TECHNIVIE
Drug: Sofosbuvir — Tablet
  Other Names: Sovaldi
Drug: Ribavirin (RBV) — Tablet
  Arms: Arm B (GT3, noncirrhotic); Arm C (GT2, noncirrhotic); Arm D (GT2, noncirrhotic); Arm E (GT3, cirrhotic)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Ombitasvir (OBV)/paritaprevir (PTV)/ritonavir (r) with sofosbuvir (SOF) with or without ribavirin (RBV) in adults with Genotype 2 Chronic Hepatitis C Virus (HCV) infection or Genotype 3 HCV infection with or without Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HCV infection prior to study enrollment.
2. Screening laboratory results from the central clinical laboratory indicating HCV genotype 2 or 3 infection only (no mixed genotype).
3. Absence OR presence of cirrhosis.
4. If cirrhotic, need to have compensated cirrhosis and absence of hepatocellular carcinoma (HCC)

Exclusion Criteria:

1. Positive screen for hepatitis B surface antigen or anti-human immunodeficiency virus antibody
2. Recent (within 6 months prior to study drug administration) history of drug or alcohol abuse.
3. Current enrollment in another clinical study, previous enrolment in this study, or previous use of any investigational or commercially available anti-HCV therapy (other than interferon, pegIFN, RBV, and or SOF) including previous exposure to telaprevir, boceprevir, ABT-450, or ombitasvir (ABT-267).
4. Subjects without cirrhosis: Any current or past clinical evidence of cirrhosis.
5. Abnormal lab tests.
6. Females who are pregnant or plan to become pregnant or breastfeeding, or males whose partners are pregnant or planning to become pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariem Charafeddine, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shafran SD, Shaw D, Charafeddine M, Agarwal K, Foster GR, Abunimeh M, Pilot-Matias T, Pothacamury RK, Fu B, Cohen E, Cohen DE, Gane E. Efficacy and safety results of patients with HCV genotype 2 or 3 infection treated with ombitasvir/paritaprevir/ritonavir and sofosbuvir with or without ribavirin (QUARTZ II-III). J Viral Hepat. 2018 Feb;25(2):118-125. doi: 10.1111/jvh.12782. Epub 2017 Sep 14. PMID 28833938
- [Derived] King JR, Dutta S, Cohen D, Podsadecki TJ, Ding B, Awni WM, Menon RM. Drug-Drug Interactions between Sofosbuvir and Ombitasvir-Paritaprevir-Ritonavir with or without Dasabuvir. Antimicrob Agents Chemother. 2015 Nov 23;60(2):855-61. doi: 10.1128/AAC.01913-15. Print 2016 Feb. PMID 26596948

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 35-day screening period.
Period: Overall Study
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic)
Started | 9 | 11 | 10 | 9 | 21 | 10
Completed | 9 | 11 | 9 | 8 | 20 | 10
Not Completed | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Subject enrolled in new study. | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study drug were included in the intent-to-treat (ITT) population; the safety population is the same as the ITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic) | Total
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 21 | 10 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (9.17) | 53.5 (8.26) | 56.6 (6.70) | 61.6 (5.90) | 53.8 (6.56) | 48.9 (7.52) | 54.2 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 3 | 9 | 2 | 27
  Male | 5 | 7 | 5 | 6 | 12 | 8 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 11 | 10 | 7 | 17 | 9 | 61
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 2 | 1 | 1 | 5
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic)
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 21 | 10
percentage of participants | 100 [70.1 to 100] | 90.9 [62.3 to 98.4] | 90.0 [59.6 to 98.2] | 44.4 [18.9 to 73.3] | 100 [84.5 to 100] | 100 [72.2 to 100]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment; confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment for 12-week and 8-week treatment or at least 26 days of treatments for 6-week treatment.
Time Frame: Up to Week 12
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic)
Number analyzed (Participants) | 9 | 11 | 10 | 9 | 21 | 10
percentage of participants | 0 [0.0 to 29.9] | 0 [0.0 to 25.9] | 0 [0.0 to 27.8] | 0 [0.0 to 29.9] | 0 [0.0 to 15.5] | 0 [0.0 to 27.8]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: Up to 12 weeks after the last actual dose of active study drug
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic)
Number analyzed (Participants) | 9 | 10 | 10 | 9 | 21 | 10
percentage of participants | 0 [0.0 to 29.9] | 0 [0.0 to 27.8] | 10.0 [1.8 to 40.4] | 55.6 [26.7 to 81.1] | 0 [0.0 to 15.5] | 0 [0.0 to 27.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks).
Description: TEAEs and and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Arm A (Genotype [GT]3, Noncirrhotic): Ombitasvir (OBV)/paritaprevir (PTV)/ritonavir (r) 25/150/100 mg once daily (QD ) and sofosbuvir (SOF) 400 mg QD for 12 weeks.
- Arm C (GT2, Noncirrhotic): OBV/PTV/r (25/150/100) mg QD with SOF (400 mg QD) and RBV (weight-based 1,000 mg or 1,200 mg daily divided BID) for 8 weeks.
Arm/Group | Arm A (Genotype [GT]3, Noncirrhotic) | Arm B (GT3, Noncirrhotic) | Arm C (GT2, Noncirrhotic) | Arm D (GT2, Noncirrhotic) | Arm E (GT3, Cirrhotic) | Arm F (GT3, Noncirrhotic)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11 | 0/10 | 0/9 | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 1/10 | 0/9 | 2/21 | 0/10
Other Adverse Events (participants affected / at risk) | 8/9 | 10/11 | 10/10 | 9/9 | 20/21 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genotype [GT]3, Noncirrhotic) (N=9) | Arm B (GT3, Noncirrhotic) (N=11) | Arm C (GT2, Noncirrhotic) (N=10) | Arm D (GT2, Noncirrhotic) (N=9) | Arm E (GT3, Cirrhotic) (N=21) | Arm F (GT3, Noncirrhotic) (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genotype [GT]3, Noncirrhotic) (N=9) | Arm B (GT3, Noncirrhotic) (N=11) | Arm C (GT2, Noncirrhotic) (N=10) | Arm D (GT2, Noncirrhotic) (N=9) | Arm E (GT3, Cirrhotic) (N=21) | Arm F (GT3, Noncirrhotic) (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (3) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 6 (10) | 3 (3)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENERGY INCREASED (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 3 (3) | 3 (4) | 6 (9) | 10 (13) | 4 (4)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 5 (5) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
POLYDIPSIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 4 (4) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 6 (8) | 3 (4) | 9 (9) | 2 (2)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POOR QUALITY SLEEP (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
TEARFULNESS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WITHDRAWAL SYNDROME (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHROMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIPPLE PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 7 (7) | 1 (1)
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SKIN ODOUR ABNORMAL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/19/NCT02292719/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT02292719/SAP_001.pdf